CLINICAL TRIAL: NCT01790087
Title: A Four Period, Four-Arm, Crossover Design, Randomized, Placebo and Active Controlled Study for the Evaluation of the Effect of Therapeutic and Supratherapeutic Single-Dose ANX-188 on the QT/QTc Intervals in Healthy Volunteers
Brief Title: ANX-188 Thorough QT/QTc Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mast Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ANX-188-05
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
MeSH Terms: interventions — Sodium Chloride; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ANX-188 Therapeutic dose level (Experimental): IV administration. 100 mg/kg for one hour followed by 30 mg/kg/hour for five hours
  Interventions: Drug: ANX-188 Therapeutic Dose
- ANX-188 Supratherapeutic dose (Experimental): IV administration. 300 mg/kg for one hour followed by 200 mg/kg/hr for five hours
  Interventions: Drug: ANX-188 Supratherapeutic dose
- Saline (Placebo Comparator): IV administration. Six hour infusion.
  Interventions: Drug: Saline
- Moxifloxacin (Active Comparator): Oral tablet. 400 mg.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: ANX-188 Therapeutic Dose
  Other Names: vepoloxamer
  Arms: ANX-188 Therapeutic dose level
Drug: ANX-188 Supratherapeutic dose
  Other Names: vepoloxamer
  Arms: ANX-188 Supratherapeutic dose
Drug: Saline
  Other Names: Placebo Comparator
  Arms: Saline
Drug: Moxifloxacin
  Other Names: Active Comparator
  Arms: Moxifloxacin

SUMMARY:
This study has been designed in compliance with the ICH-E14 guideline (2005) to evaluate the effect of ANX-188 at therapeutic and supratherapeutic concentrations on cardiac repolarization, specifically, Fridericia's QT-Interval (QTcF)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18 to 65 (inclusive) in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory testing at screening.

Exclusion Criteria:

* Participation in a clinical trial within the last 60 days
* Pregnant or lactating females
* Use of prescription drugs, herbals, or over-the-counter medications within 14 days prior to study day -2
* Uncontrolled cardiac arrhythmias, cardiac valve abnormalities, or not in normal sinus rhythm
* Smokers or tobacco product user in the prior 3 months
* Presence of clinically significant illness
* Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of therapeutic and supratherapeutic doses of ANX-188 on cardiac ventricular repolarization, specifically, the Fridericia's corrected QT-Interval (QTcF) | Day 1 Pre-dose to 24 hours post-dose

SECONDARY OUTCOMES:
Bazett's corrected QT-interval (QTcB) | Pre-dose to 24 hours post-dose
Heart rate measurements on treatment compared to time-matched baseline and placebo | Pre-dose to 24 hours post-dose
RR-interval on treatment compared to time-matched baseline and placebo | Pre-dose to 24 hours post-dose
QRS measurements on treatment compared to time-matched baseline and placebo | Pre-dose to 24 hours post-dose
PR interval measurements on treatment compared to time-matched baseline and placebo | Pre-dose to 24 hours post-dose
Overall characterization of normal and abnormal ECGs and the number and percentage of subjects with normal and abnormal ECGs | Pre-dose to 24 hours post-dose
Number and percentage of subjects that develop abnormalities of repolarization on treatment | Pre-dose to 24 hours post-dose
Number and percentage of subjects the develop abnormal U waves | Pre-dose to 24 hours post-dose
Relationship between changes from the baseline and placebo in QTcF (DDQTcF) | Pre-dose to 24 hours post-dose
Analysis for arrhythmias | Pre-dose to 24 hours post-dsoe
Correlation of ECG findings with clinical adverse events | Pre-dose to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Edwin L Parsley, D.O., Study Director — Mast Therapeutics
Locations (1):
- Research Site, Baltimore, Maryland, United States